CLINICAL TRIAL: NCT06129799
Title: Exercise CMR in (Paradoxical) Low-flow Low-gradient Aortic Stenosis
Brief Title: Exercise CMR in (p)LF-LG AS
Status: Recruiting | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Sören Backhaus, Principal Investigator, University of Göttingen
Other Study IDs: 16822
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- paradoxical LF-LG AS
- conventional LF-LG AS

SUMMARY:
Patient with paradoxical or conventional low-flow low-gradient aortic stenosis on echocardiographic assessment will undergo physiological exercise-stress CMR in addition to guideline recommended surveys prior to TAVR.

ELIGIBILITY:
Inclusion Criteria:

* paradoxical or conventional severe low-flow low-gradient aortic stenosis

Exclusion Criteria:

* CMR incapable device
* unable to undergo 40 min scan (can not lie flat, claustrophobia)
* renal insufficiency (eGFR <30 ml/min/1.73m²)
* allergy against contrast agent
* unable to exercise in supine position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prior to TAVR
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of events: number of participants with cardiovascular death or heart failure hospitalisation | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Goettingen, Göttingen, Germany